CLINICAL TRIAL: NCT01348841
Title: Wound Interdisciplinary Teams (WIT): A Community- Based Pragmatic Randomized Controlled Trial
Acronym: WIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Murray Krahn, Director, THETA, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 25973
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Wound of Skin
Keywords: community wound care; systematic wound team referral; Advanced in-home nurse wound training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (No Intervention): Usual care is care as currently delivered to clients with chronic wounds in the community.
- Intervention Arm (Experimental): Systematic referral to MDWCT and comprehensive primary care:
  Intervention consists of systematic referral to MDWCT in conjunction with comprehensive primary care.Systematic referral to, and follow up, by MDWCTs, co-ordinated by the CM, will occur.There will be immediate referral to the MDWCT of clients with :1/ diabetic lower extremity ulcers,2/peripheral neuropathy, charcot changes,3/wound present longer than 4 mths. ,4/ Ankle Brachial Index less than 0.6, non-diabetics, and not being seen by a vascular surgeon. Subsequent referral to MDWCT will occur if less than 30% healing by week 4.
  Interventions: Other: Systematic referral to MDWCT and comprehensive primary care

INTERVENTIONS:
Other: Systematic referral to MDWCT and comprehensive primary care — Systematic referral to, and follow up, by Multi-Disciplinary Wound Care Teams (MDWCTs), co-ordinated by the Case Manager (CM), will occur.There will be immediate referral to the MDWCT of clients with :1/ diabetic lower extremity ulcers,2/peripheral neuropathy, charcot changes,3/wound present longer than 4 mths. ,4/ Ankle Brachial Index less than 0.6, non-diabetics, and not being seen by a vascular surgeon. Subsequent referral to MDWCT will occur if less than 30% healing by week 4.
  Other Names: systematic expedited referral to MDWCTs
  Arms: Intervention Arm

SUMMARY:
Wounds that are slow to heal (chronic) may be managed in different ways. In Ontario, care in the community for most of these is coordinated by the local Community Care Access Centre (CCAC). One or more health professionals might deliver treatment, individually or as part of a wound care team, with different members having different kinds of training (interdisciplinary team), which may or may not include wound care. Community treatment by interdisciplinary teams has been shown to be more effective and cost-effective for some long-standing health problems, but further scientific evidence is needed to determine if this is also true for chronic wounds.

This study compares the usual way chronic wounds are being managed in the community with a so-called "intermediate care" approach. In this study, intermediate care will involve health service providers following certain agreed-upon steps (evidence-based best practice) from first contact with the client through assessment, treatment, and on to referral to a hospital specialty wound care team, if needed.

DETAILED DESCRIPTION:
For certain types of chronic illness, planning case management and providing care according to evidence-based guidelines (published methods that have been supported scientifically) results in better clinical outcomes and better cost-effectiveness. Wound management by interdisciplinary teams may have these advantages in both the community primary care setting and the hospital specialized care setting. Systematic review of the literature indicated that the evidence was incomplete to support implementation of an intermediate care model for community management of chronic wounds. Therefore, the Ontario Health Technology Advisory Committee recommended that a field evaluation be conducted to provide stronger evidence about the relative effectiveness, cost-effectiveness and feasibility of managing chronic wounds in the community using both standardized, comprehensive primary care and a systematic method of referral to a specialty, multidisciplinary team based in a hospital

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years of age) client with eligible wound type (not surgical, malignant or burns) referred to the Toronto Central CCAC for wound management.
* Client (or substitute decision maker) provides written, informed consent.
* Someone in client's home (or substitute decision maker) must be able to speak English.

Exclusion Criteria:

* Surgical wounds
* Burns
* Malignant wounds
* Clients who are designated palliative on CCAC referral form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Time to Healing | 6 months
  The primary clinical outcome measure will be time to healing, ascertained by digital wound photography using computer planimetry for wound measurement.

SECONDARY OUTCOMES:
proportion of wound healed | 6 months
  proportion of wounds healed at 6 mths and the rate of wound healing(cm2/week).
Wound recurrence | 6 months
  Wound recurrence within the study period.
time to discontinuation of wound service | 1 years
  Time to discontinuation of wound services within the CCAC and interdisciplinary teams.
Health Related Quality of Life (HRQOL) | 6 months
  Health related quality of life.
client satisfaction | 6 months
  Satisfaction with care.
cost and resource use | 6 months
  cost and resource use of wound care provided

CONTACTS AND LOCATIONS:
Overall Officials: Murray Krahn, PhD, MD, Principal Investigator — Director
Locations (1):
- THETA Collaborative, Toronto, Ontario, Canada

REFERENCES:
- [Background] Bennett G, Dealey C, Posnett J. The cost of pressure ulcers in the UK. Age Ageing. 2004 May;33(3):230-5. doi: 10.1093/ageing/afh086. PMID 15082426
- [Background] Xakellis GC, Frantz R. The cost of healing pressure ulcers across multiple health care settings. Adv Wound Care. 1996 Nov-Dec;9(6):18-22. PMID 9069752
- [Background] Watson JM, Kang'ombe AR, Soares MO, Chuang LH, Worthy G, Bland JM, Iglesias C, Cullum N, Torgerson D, Nelson EA; VenUS III team. VenUS III: a randomised controlled trial of therapeutic ultrasound in the management of venous leg ulcers. Health Technol Assess. 2011 Mar;15(13):1-192. doi: 10.3310/hta15130. PMID 21375959
- [Background] Jeffcoate WJ, Price PE, Phillips CJ, Game FL, Mudge E, Davies S, Amery CM, Edmonds ME, Gibby OM, Johnson AB, Jones GR, Masson E, Patmore JE, Price D, Rayman G, Harding KG. Randomised controlled trial of the use of three dressing preparations in the management of chronic ulceration of the foot in diabetes. Health Technol Assess. 2009 Nov;13(54):1-86, iii-iv. doi: 10.3310/hta13540. PMID 19922726
- [Background] Hawes C, Fries BE, James ML, Guihan M. Prospects and pitfalls: use of the RAI-HC assessment by the Department of Veterans Affairs for home care clients. Gerontologist. 2007 Jun;47(3):378-87. doi: 10.1093/geront/47.3.378. PMID 17565102
- [Background] Fries BE, James M, Hammer SS, Shugarman LR, Morris JN. Is telephone screening feasible? Accuracy and cost-effectiveness of identifying people medically eligible for home- and community-based services. Gerontologist. 2004 Oct;44(5):680-8. doi: 10.1093/geront/44.5.680. PMID 15498843
- [Background] Torrance GW, Furlong W, Feeny D, Boyle M. Multi-attribute preference functions. Health Utilities Index. Pharmacoeconomics. 1995 Jun;7(6):503-20. doi: 10.2165/00019053-199507060-00005. PMID 10155336
- [Background] Wodchis WP, Hirdes JP, Feeny DH. Health-related quality of life measure based on the minimum data set. Int J Technol Assess Health Care. 2003 Summer;19(3):490-506. doi: 10.1017/s0266462303000424. PMID 12962335
- [Background] Wodchis WP, Maxwell CJ, Venturini A, Walker JD, Zhang J, Hogan DB, Feeny DF. Study of observed and self-reported HRQL in older frail adults found group-level congruence and individual-level differences. J Clin Epidemiol. 2007 May;60(5):502-11. doi: 10.1016/j.jclinepi.2006.08.009. Epub 2007 Jan 18. PMID 17419961
- [Background] Burrows AB, Morris JN, Simon SE, Hirdes JP, Phillips C. Development of a minimum data set-based depression rating scale for use in nursing homes. Age Ageing. 2000 Mar;29(2):165-72. doi: 10.1093/ageing/29.2.165. PMID 10791452